CLINICAL TRIAL: NCT04395625
Title: Computer-aided Indirect Bonding Versus Traditional Direct Bonding of Brackets in Orthodontic Patients: a Randomized Controlled Trial
Brief Title: Computer-aided Indirect Bonding Versus Traditional Direct Bonding of Brackets in Orthodontic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10101
Record Dates: First submitted 2020-05-05; First posted 2020-05-20 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Orthodontic Appliances, Fixed
Keywords: Indirect bonding; CAD/CAM; Time; Cost-minimization analysis; Failure rate

STUDY DESIGN:
Intervention Model Description: Single-center 2-arm parallel randomized controlled trial with a 1:1 allocation ratio, following a split-mouth design.
Who Masked: Outcomes Assessor
Masking Description: During data analysis, anonymization is ensured by assigning a number to each patient, so that the investigator is blinded to the patient's group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Patients had their upper right and lower left quadrants bonded with indirect bonding, and their upper left and lower right quadrants with direct bonding.
  Interventions: Procedure: Direct bonding of Orthodontic brackets; Procedure: Indirect bonding of Orthodontic brackets
- Group 2 (Experimental): Patients had their upper left and lower right quadrants bonded with indirect bonding, and their upper right and lower left quadrants with direct bonding.
  Interventions: Procedure: Direct bonding of Orthodontic brackets; Procedure: Indirect bonding of Orthodontic brackets

INTERVENTIONS:
Procedure: Direct bonding of Orthodontic brackets — Patients in group 1 had their upper right and lower left quadrants bonded with indirect bonding, and their upper left and lower right quadrants with direct bonding
Procedure: Indirect bonding of Orthodontic brackets — Patients in group 2 had their upper left and lower right quadrants bonded with indirect bonding, and their upper right and lower left quadrants with direct bonding.

SUMMARY:
Accurate bracket positioning is one of the keys for effective orthodontic treatment. Traditionally, orthodontic brackets are positioned one-by-one on the teeth of the patient, with the so-called direct bonding method.

In the past, the term indirect bonding defined a technique where the brackets were positioned on a plaster model in order to increase placement precision. A transfer tray was then built on the plaster, incorporating all the brackets mounted. Finally, this transfer tray was positioned in the mouth of the patient, so that all the brackets could be bonded to the teeth at once in the pre-determined position. Several studies have investigated this indirect technique based on plaster models.

With computer-aided technology, a new form of digital indirect bonding is now possible. The dentist digitally places the brackets on a virtual 3D model of the teeth. A tray with the brackets' positioning information is then generated with CAD-CAM (computer aided design and manufacturing) technology and the brackets are subsequently indirectly transferred to the teeth. This new approach could possibly save chair time and increase precision. Our profession is today moving towards the virtual reality, and application of such a computer-aided technology method into the clinical work-flow seems definitely promising for our future daily practice.

Since the evidence about this new computer-assisted indirect bracket bonding method is very limited, the purpose of this study is to evaluate precision, chair time, and bracket survival by comparing this digital indirect bonding method to the traditional direct bonding method

Specific objectives

* To assess and compare the accuracy of a conventional direct bonding method with an indirect computer-aided bonding method.
* To evaluate chair time and bracket survival related to both bonding methods.

Hypothesis

Null hypothesis:

I. There is no difference in accuracy of bracket placement between the direct and indirect bonding methods.

II. There is no difference in chair time between the two bonding methods. III. Bracket bond failure is similar for both bonding methods.

Alternative hypothesis:

I. Bracket placement is more precise/accurate with the indirect bonding method compared to the traditional direct bonding method.

II. Indirect bonding reduces chair time.

DETAILED DESCRIPTION:
Trial design:

2-arm parallel randomized clinical trial.

Participants, eligibility criteria and settings:

Consecutive patients seeking orthodontic treatment at the Section of Orthodontics, School of Dentistry, Aarhus University, previously selected to be suitable for full fixed appliance with metallic brackets in the Postgraduate clinic, according to treatment needs.

The following inclusion criteria will be applied: minimum 4 permanent teeth (except molars) to be bonded in each of the 4 quadrants (thus extraction or non-extraction cases) and with all teeth fully erupted.

Exclusion criteria: presence of active caries, fluorosis or hypoplasia of enamel, restorations or fractures of the surfaces to be bonded, abnormalities in crown morphology of teeth to be bonded. Subject with major rotations impeding proper bracket positioning will also be excluded.

The patients will be informed about the study orally and in a written form. Consent from patients or parents (if the patient is adolescent) will be obtained before the bonding procedure.

Sample size:

According to the literature, failure of brackets is varying from 3 to 30% [9, 10]. Calculation of sample size for determination of equivalence of 2 proportions (expected proportion of failures in control group: 25% - expected proportion of failures in test group: 25% - maximum permitted difference: 10%) resulted in a sample size of 232 brackets per group, for a p=0.05 and a power of 80%. This corresponds to 29 patients (232/8). A sample size of 40 patients will be used in order to account for potential drop-outs.

Randomization:

Subjects will be randomly allocated into one of two groups with a different split mouth set-up (Table). Randomization with a 1:1 allocation using random block size of 4 will be applied, following a sequence generated online (randomization.com). Allocation to groups will take place before laboratory ordering. Allocation concealment will be ensured by using sealed envelopes.

Intervention-Protocol:

Treatment will be performed by postgraduate students (hereinafter referred to as "dentist") in the Postgraduate clinic at the Section of Orthodontics (School of Dentistry, Aarhus University). All patients will have metallic brackets bonded from 2nd premolar to 2nd premolar.

1. Impression and laboratory procedure:

   1. Alginate impression;
   2. Laboratory work : impression will be poured and plaster model will be scanned creating digital models of the malocclusion of the patient;
   3. The digital model will be imported in the software . Here the dentist will digitally place the brackets on the teeth of the two quadrants selected for indirect bonding according to randomization (Group 1 or Group 2);
   4. Laboratory work : two individual bonding trays (one per quadrant) made of a rigid-elastic plastic material will be produced by CAD-CAM, following the brackets positioning information as predefined by the dentist. The actualbrackets will thus be engaged in the bonding trays. The trays hosting the brackets will be delivered to the clinic, ready to be used by the dentist.
2. Bonding procedures:

   A cheek retractor will be placed. The buccal surface of all teeth from premolar to premolar will be pumiced, then acid-etched with 37% phosphoric acid (30s), rinsed and dried. The two quadrants allocated to indirect bonding will be bonded first. Bonding of the two remaining quadrant using the direct bonding method will be done in second instance.
   1. Indirect bonding method:

      The trays will be tried in the mouth. If they can be inserted at once, this will be preferred. If insertion in one piece is not possible, the tray will be fractioned in 2 or more pieces. The etched enamel surface of the teeth in the two quadrants selected for indirect bonding will be prepared with adhesive . The base of all brackets engaged in the first tray will be covered with a thin layer of light cure composite for bonding. This tray with the brackets will subsequently be placed on the teeth. The dentist will remove the excess of composite and then light cure for 10 seconds per bracket with a polymerization light . After light-curing, the tray will be cut with a carbide bur and will be removed from the mouth of patient. This operation will be repeated for the second tray.
   2. Direct bonding method:

   The etched enamel surface of the teeth in the two quadrants selected for direct bonding will be prepared with adhesive and brackets will be positioned one-by-one by the dentist, using bracket tweezers and height gauges, after coating the bracket base with light cure composite. The dentist will remove the excess of composite and then light-cure for 10 seconds per bracket with a polymerization light.

   The time for bonding with each method will be recorded (in seconds) with a timer.

   After bonding all quadrants, in case of presence of premature contacts on the brackets, the bite will be raised with bite blocks.

   Wires will be engaged and potential immediate debondings will be recorded. If extractions are part of the treatment plan, these extractions will be postponed after bonding.

   All patients will be informed about hygiene and diet recommendations.
3. Follow-up during orthodontic treatment:

   1. Bracket bonding failure (type of tooth and type of failure - i.e. at the bracket-composite or at the composite-enamel interface -) will be recorded at every orthodontic visit (every 4 to 6 weeks), until debonding at the end of treatment (approximately 18-36 months later);
   2. Six to twelve months after bonding as well as at the end of treatment, bracket position accuracy will be evaluated on digital models produced by intraoral scanning;
   3. In accordance with the standard orthodontic treatment protocol in the Postgraduate clinic at the Section of Orthodontics, a panoramic radiograph will be taken 6 to 12 months after bonding as well as at the end of treatment in order to assess the influence of brackets placement on the position of the teeth and roots;
   4. Finally, the number of brackets rebonded as well as the number of finishing bends, which are needed because of unsatisfactory bracket positioning, will be recorded at every orthodontic visit (every 4 to 6 weeks), until end of treatment.
4. Follow-up after treatment:

Patients will be recalled 2 and 5 years after the end of treatment. Treatment stability will be assessed on digital models produced by intraoral scanning.

Statistical analysis:

Collected data will be anonymized and analyzed in a blinded way. All analyses will be conducted using SPPS statistic software.

Information regarding sex, age and malocclusion (e.g. Angle classification) will be analyzed with descriptive statistics.

Paired t-tests will be used to compare bonding time between the two methods, after checking for normality.

The log-rank test will be used to compare the Kaplan Meier survival curves of the two methods. A test of proportion will be applied to compare the failures at different time points between bonding methods.

Accuracy will be evaluated by scoring bracket positioning both on digital models and panoramic radiographs for every tooth, at all time-points. Kappa statistics will be used to compare the scores.

Descriptive statistics will be used to describe long term stability.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients selected to be suitable for full fixed appliance according to treatment needs and accepting to have metallic brackets.
* Presence of minimum four permanent teeth (except molars) to be bonded in each of the 4 quadrants (thus extraction or non-extraction cases)
* All teeth fully erupted.

Exclusion Criteria:

* Patients with teeth presenting active caries, fluorosis or hypoplasia of enamel, restorations or fractures of the surfaces to be bonded, or abnormalities in crown morphology of the teeth to be bonded.
* Subjects with major rotations impeding proper bracket positioning.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Time | On the day the brackets are bonded (bonding date): within 24 hours
  Time used for bonding brackets with the CAD/CAM indirect and the traditional direct bonding techniques

SECONDARY OUTCOMES:
Immediate bracket failure rate | On the day the brackets are bonded (bonding date): within 24 hours
  Immediate bracket failure rate
Cost-minimization analysis | On the day the brackets are bonded (bonding date): within 24 hours
  Cost-minimization analysis
Overall bracket failure rate | From the day the brackets are bonded (bonding date) to the day the brackets are removed (debonding date), generally about 2 years later.
  Bracket failure rate throughout orthodontic treatment
Bracket position accuracy according to position of the teeth | From the day the brackets are bonded (bonding date) to the day the brackets are removed (debonding date), generally about 2 years later.
  Bracket position accuracy according to position of the teeth on intra-oral scanning
Bracket position accuracy according to axes of the roots | From the day the brackets are bonded (bonding date) to the day the brackets are removed (debonding date), generally about 2 years later.
  Bracket position accuracy according to axes of the roots on panoramic X-rays
Bracket position accuracy according to finishing bends | From the day the brackets are bonded (bonding date) to the day the brackets are removed (debonding date), generally about 2 years later.
  Bracket position accuracy according to number of finishing bends
Bracket position accuracy according to number of brackets rebonded | From the day the brackets are bonded (bonding date) to the day the brackets are removed (debonding date), generally about 2 years later.
  Bracket position accuracy according to number of brackets rebonded because of unsatisfactory bracket positioning

IPD SHARING:
Plan to Share IPD: No